CLINICAL TRIAL: NCT02403336
Title: Health Education in Perimenopausal Women to Promote Self-care and Quality of Life: Randomized Clinical Trial
Brief Title: Health Education in Perimenopausal Women to Promote Self-care and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government); Fondo de Investigacion Sanitaria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI/1100693
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Perimenopausal Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral group intervention (Experimental): Professionals: 3 training sessions for updating the knowledge and learning skills. Patients: Health education workshop.
  Interventions: Other: Training health professionals; Behavioral: Behavioral group intervention
- Usual clinical practice (Active Comparator): Professionals: meeting methodological of 30 minutes duration. Patients: Usual clinical practice. Health education individually on nursing consultation.
  Interventions: Other: Usual clinical practice

INTERVENTIONS:
Other: Training health professionals — Intervention on the professionals (3 training sessions for updating the knowledge and learning skills) and
  Arms: Behavioral group intervention
Behavioral: Behavioral group intervention — Intervention on patients (educational workshop).
  Arms: Behavioral group intervention
Other: Usual clinical practice — Professionals: meeting methodological of 30 minutes duration. Patients: Usual clinical practice. Health education individually on nursing consultation.
  Arms: Usual clinical practice

SUMMARY:
Objective: To evaluate the efficiency of a group intervention opposite to the usual care to improve the quality of life, measured with the SF-12 questionnaire, in women between 45-55 years to the primary health care centres.

DETAILED DESCRIPTION:
Methods: clinical controlled trial with parallel groups, random assignment of primary care units and blinded evaluation of principal label.

Setting: study in primary health care centres (PHCCs) of Madrid Health Service and Castilla León Health Service.

Subjects: Women between 45-55 years to medical consultation in primary care. Intervention: application of good clinical practice procedure and cognitive - behavioural grupal intervention.

Sample size: N=355 patients. Data: Principal response variables: quality of life measured with the SF-12 questionnaire. Secondary response Variables: visits number, medicine /month number, and transitory disability days. Other prognosis and descriptive variables.

Data analysis: Main effectiveness will be analyzed by comparing the improvement in 4 or more points in the SF-12 Mental Health area at 6, 12, 18 y 24 months post- intervention, between intervention and control group. Logistic regression will be used to adjust for prognostic factors. Confounding factors or factors that might alter the effect, recorder will be taken in account in this analysis. All statistical tests will be performed with intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* 45-55 years women
* users of the Health Center
* able to follow the demands of the study: does not have the intention to move from home in the next 24 months
* have ability to read and write the Spanish language and agreeing to participate by giving their informed consent in writing.

Exclusion Criteria:

* Women immobilized at home, with mental disorder or cognitive impairment and/or sensory impairments that prevent to participate in a group intervention.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 356 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 24 months
  SF-12 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Lorena LOPEZ-CASTAÑON, Moralzarzal, Madrid, Spain